CLINICAL TRIAL: NCT04896255
Title: Long-term Outcomes of Anti-viral Therapies in Patients With Chronic Viral Hepatitis B: A Multicenter, Real-world Study
Brief Title: Long-term Outcomes of Anti-viral Therapies in Patients With Chronic Viral Hepatitis B
Acronym: OASIS
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Chinese Foundation for Hepatitis Prevention and Control (Unknown); The Third People's Hospital of Taiyuan (Other); First Affiliated Hospital of Chongqing Medical University (Other); Beijing YouAn Hospital (Other); Henan Provincial People's Hospital (Other); Yunnan Provincial No.1 Hospital (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Beijing Ditan Hospital (Other); Tianjing No.2 People's Hospital (Unknown); Qingdao No.6 People's Hospital (Unknown); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Ningbo Beilun District Traditional Chinese Medicine Hospital (Other); Wuxi No.5 People's Hospital (Unknown); Taicang No.1 People's hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Other Study IDs: KY2020-911
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective: CHB patients enrolled pre-Protocol v3.0 (Dec 2023), planned or on antiviral therapy, followed prospectively for 5 years post-consent. Treatments: routine NA monotherapy, or PegIFN based regimens, per clinical guidelines. Data: baseline and 5 -year follow-up via routine visits.
  Interventions: Drug: peginterferon alpha based regimen; Drug: nucleos(t)ide
- Retrospective-Prospective: CHB patients with baseline (≥Sep 2020) pre-v3.0, consenting post-v3.0. Retrospective data from baseline to consent; prospective for 5 years from baseline. Treatments: NAs monotherapy, or PegIFN based regimens. Data: retrospective before consent; prospective from visit matching baseline-consent interval. Missing routine data noted.
  Interventions: Drug: peginterferon alpha based regimen; Drug: nucleos(t)ide
- Retrospective: CHB patients with records from Sep 2020 to v3.0 (Dec 2023), collected retrospectively. Treatments: NAs monotherapy, or PegIFN based regimens, per historical practice. Data: extracted from the electronic healthcare record; missing routine data recorded.
  Interventions: Drug: peginterferon alpha based regimen; Drug: nucleos(t)ide

INTERVENTIONS:
Drug: peginterferon alpha based regimen — peginterferon alpha based regimen or nucleos(t)ide alone are decided by patients' doctors according to their conditions, instead of extra interventions brought by the study
Drug: nucleos(t)ide — peginterferon alpha based regimen or nucleos(t)ide alone are decided by patients' doctors according to their conditions, instead of extra interventions brought by the study

SUMMARY:
The goal of this observational, multicenter , real-world study is to evaluate the long-term outcomes of different antiviral therapies in adults with chronic hepatitis B (CHB). The main questions it aims to answer are: What is the 5-year incidence of hepatocellular carcinoma (HCC) under various treatment regimens? How do rates of HBsAg seroclearance, decompensated cirrhosis, liver fibrosis progression, and other virological and clinical outcomes compare across regimens? Researchers will compare real-world treatment arms-including nucleos(t)ide analogue (NA) monotherapy (e.g., entecavir, tenofovir), PegIFN based regimen (e.g., PegIFN monotherapy, PegIFN plus NA combinations)-to identify optimal strategies for reducing HCC risk and improving functional cure rates.

Participants will undergo routine clinical care with no study-imposed interventions; data on demographics, medical history, symptoms, laboratory tests (e.g., HBsAg, HBV DNA, liver function), imaging (e.g., ultrasound, elastography), and clinical events will be collected prospectively (for up to 5 years in some cohorts) or retrospectively from medical records at baseline and scheduled follow-up visits (e.g., every 3-12 months initially, then annually).

DETAILED DESCRIPTION:
The OASIS study is a multicenter, observational, real-world cohort study designed to evaluate long-term outcomes of antiviral therapies for chronic hepatitis B (CHB). It compares nucleos(t)ide analogue (NA) monotherapy, pegylated interferon based regimen without randomization or blinding. Treatment decisions follow routine clinical guidelines, physician expertise, and patient-specific factors. The study includes three cohorts: Prospective (PS, 5-year follow-up post-consent), Retrospective-Prospective (RPS, retrospective from baseline ≥September 2020 to consent, then 5-year prospective), and Retrospective (RS, data from September 2020 to protocol implementation). The target of 33,000 patients was determined based on patient flow across sub-centers, ensuring sufficient power to detect differences in 5-year HCC incidence (primary endpoint) and secondary outcomes (e.g., HBsAg seroclearance rates).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age ≥18; subjects who are over 70 years of age must be in generally stable health conditions.
* There should be evidences that HBsAg has been positive for more than 6 months or HBV-related histological changes.
* Planned or currently receiving potent low-resistance NAs [entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), or tenofovir amibufenamide (TMF)], or planned to receive PegIFNα-2b, either treated or treatment-naïve.
* Agree to participate in the study and sign the patient informed consent form.

Exclusion Criteria:

* Hepatocellular carcinoma (diagnosed or planned for treatment) or liver failure at baseline
* Concurrently participating in other interventional clinical trials.
* Any other conditions deemed unsuitable by investigators or preventing compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hepatitis B under anti-viral treatment of peginterferon alpha based regimen or nucleos(t)ide alone.
Sampling Method: Non-Probability Sample
Enrollment: 33000 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of hepatocellular carcinoma at 5 year from baseline | 5 year from baseline
  Rate of hepatocellular carcinoma will be evaluated as an end-stage liver disease event at 5 years from baseline

SECONDARY OUTCOMES:
rate of HBsAg loss | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  rate of HBsAg loss will be measured as a serological response event at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively.
rate of decompensated cirrhosis | 1year, 2 year, 3 year, 4 year and 5 year from baseline
  Rate of decompensated cirrhosis will be evaluated as an end-stage liver disease event at 1year, 2 year, 3 year, 4 year, and 5 year from baseline
rate of cirrhosis | 1 year, 2 year, 3 year, 4year, and 5 year from baseline
  rate of cirrhosis at 1 year, 2 year, 3 year, 4year, and 5 year from baseline
rate of fibrosis progression | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  rate of fibrosis progression will be measured as a histological response event at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively.
rate of fibrosis regression | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  rate of fibrosis regression will be measured as a histological response event at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively.
rate of liver transplantation | 5 year from baseline
  Rate of liver transplantation will be evaluated as an end-stage liver disease event at 5 year from baseline
HBsAg level | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  HBsAg level will be measured at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively, and kinetics will be described based on the results.
rate of HBeAg loss | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  rate of HBeAg loss will be measured as a serological response event at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively.
rate of HBeAg conversion | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline
  rate of HBeAg conversion will be measured as a serological response event at 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 168 weeks, 192 weeks, 216 weeks, 240 weeks from baseline, respectively.
rate of HBV DNA undetectable | 1year, 2 year, 3 year, 4 year and 5 year from baseline
  Rate of HBV DNA undetectable will be evaluated as an end-stage liver disease event at 1year, 2 year, 3 year, 4 year, and 5 year from baseline

OTHER OUTCOMES:
demographic characteristics | baseline
  demographic characteristics at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, MD, Principal Investigator — Huashan Hospital; Jiming Zhang, MD, Principal Investigator — Huashan Hospital; Feng Sun, MD, Study Chair — Huashan Hospital; Qiran Zhang, MD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

REFERENCES:
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Shin EC, Sung PS, Park SH. Immune responses and immunopathology in acute and chronic viral hepatitis. Nat Rev Immunol. 2016 Aug;16(8):509-23. doi: 10.1038/nri.2016.69. Epub 2016 Jul 4. PMID 27374637
- [Background] Nassal M. HBV cccDNA: viral persistence reservoir and key obstacle for a cure of chronic hepatitis B. Gut. 2015 Dec;64(12):1972-84. doi: 10.1136/gutjnl-2015-309809. Epub 2015 Jun 5. PMID 26048673
- [Background] Tang LSY, Covert E, Wilson E, Kottilil S. Chronic Hepatitis B Infection: A Review. JAMA. 2018 May 1;319(17):1802-1813. doi: 10.1001/jama.2018.3795. PMID 29715359
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on Prevention, Diagnosis, and Treatment of Chronic Hepatitis B: AASLD 2018 Hepatitis B Guidance. Clin Liver Dis (Hoboken). 2018 Aug 22;12(1):33-34. doi: 10.1002/cld.728. eCollection 2018 Jul. No abstract available. PMID 30988907
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Lim TH, Gane E, Moyes C, Borman B, Cunningham C. HBsAg loss in a New Zealand community study with 28-year follow-up: rates, predictors and long-term outcomes. Hepatol Int. 2016 Sep;10(5):829-37. doi: 10.1007/s12072-016-9709-6. Epub 2016 Mar 8. PMID 26957439
- [Background] Hu P, Shang J, Zhang W, Gong G, Li Y, Chen X, Jiang J, Xie Q, Dou X, Sun Y, Li Y, Liu Y, Liu G, Mao D, Chi X, Tang H, Li X, Xie Y, Chen X, Jiang J, Zhao P, Hou J, Gao Z, Fan H, Ding J, Zhang D, Ren H. HBsAg Loss with Peg-interferon Alfa-2a in Hepatitis B Patients with Partial Response to Nucleos(t)ide Analog: New Switch Study. J Clin Transl Hepatol. 2018 Mar 28;6(1):25-34. doi: 10.14218/JCTH.2017.00072. Epub 2018 Mar 17. PMID 29577029
- [Background] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Background] Mak LY, Wong DK, Pollicino T, Raimondo G, Hollinger FB, Yuen MF. Occult hepatitis B infection and hepatocellular carcinoma: Epidemiology, virology, hepatocarcinogenesis and clinical significance. J Hepatol. 2020 Oct;73(4):952-964. doi: 10.1016/j.jhep.2020.05.042. Epub 2020 Jun 3. PMID 32504662
- [Background] Shiels MS, Engels EA, Yanik EL, McGlynn KA, Pfeiffer RM, O'Brien TR. Incidence of hepatocellular carcinoma among older Americans attributable to hepatitis C and hepatitis B: 2001 through 2013. Cancer. 2019 Aug 1;125(15):2621-2630. doi: 10.1002/cncr.32129. Epub 2019 Apr 12. PMID 30980394
- [Background] Hsu YC, Wong GL, Chen CH, Peng CY, Yeh ML, Cheung KS, Toyoda H, Huang CF, Trinh H, Xie Q, Enomoto M, Liu L, Yasuda S, Tanaka Y, Kozuka R, Tsai PC, Huang YT, Wong C, Huang R, Jang TY, Hoang J, Yang HI, Li J, Lee DH, Takahashi H, Zhang JQ, Ogawa E, Zhao C, Liu C, Furusyo N, Eguchi Y, Wong C, Wu C, Kumada T, Yuen MF, Yu ML, Nguyen MH. Tenofovir Versus Entecavir for Hepatocellular Carcinoma Prevention in an International Consortium of Chronic Hepatitis B. Am J Gastroenterol. 2020 Feb;115(2):271-280. doi: 10.14309/ajg.0000000000000428. PMID 31634265
- [Background] Miyake Y, Kobashi H, Yamamoto K. Meta-analysis: the effect of interferon on development of hepatocellular carcinoma in patients with chronic hepatitis B virus infection. J Gastroenterol. 2009;44(5):470-5. doi: 10.1007/s00535-009-0024-z. Epub 2009 Mar 25. PMID 19308310
- [Background] Shiffman ML. Approach to the patient with chronic hepatitis B and decompensated cirrhosis. Liver Int. 2020 Feb;40 Suppl 1:22-26. doi: 10.1111/liv.14359. PMID 32077612
- [Background] Jang JW, Choi JY, Kim YS, Yoo JJ, Woo HY, Choi SK, Jun CH, Lee CH, Sohn JH, Tak WY, Lee YR, Han KH. Effects of Virologic Response to Treatment on Short- and Long-term Outcomes of Patients With Chronic Hepatitis B Virus Infection and Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2018 Dec;16(12):1954-1963.e3. doi: 10.1016/j.cgh.2018.04.063. Epub 2018 May 9. PMID 29753085

DOCUMENTS (1):
  • Study Protocol (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT04896255/Prot_000.pdf